CLINICAL TRIAL: NCT03747055
Title: Effectiveness of Group Focused Psychosocial Support to Improve the Psychosocial Well-being and Functioning of Adults Affected by Humanitarian Crisis in Nepal
Brief Title: Effectiveness of Group Focused Psychosocial Support for Adults Affected by Humanitarian Crises
Acronym: GroupPM+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: World Health Organization (Other); Transcultural Psychosocial Organization Nepal (Other); Duke University (Other); King's College London (Other)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Associate Professor of Psychiatry, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERC.0002817 Group PM+
Record Dates: First submitted 2018-10-31; First posted 2018-11-20 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Depression; Posttraumatic Stress Disorder; Psychological Distress
Keywords: Nepal; Psychological treatment; Task shifting; Humanitarian crisis
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group problem management plus (Experimental): Five sessions of group low intensity psychological intervention
  Interventions: Behavioral: Group problem management plus
- Enhanced treatment as usual (Active Comparator): Referral to primary health care workers trained in mental health Gap Action Programme.
  Interventions: Behavioral: Enhanced treatment as usual

INTERVENTIONS:
Behavioral: Group problem management plus — Low intensity group psychological intervention including stress management, behavioral activation, problem solving, and strengthening social support
  Arms: Group problem management plus
Behavioral: Enhanced treatment as usual — Referral to primary care workers trained in mental health Gap Action Program Implementation Guide
  Other Names: mental health Gap Action Program-Implementation Guide
  Arms: Enhanced treatment as usual

SUMMARY:
This is an effectiveness study of group problem management plus, a low-intensity psychological intervention, delivered in five sessions to adults affected by humanitarian crises. The current study will evaluate the effectiveness of Group Problem Management Plus (PM+).

DETAILED DESCRIPTION:
Counselling programmes used in many humanitarian settings are often non- specific with unknown efficacy and safety. Only a few interventions in humanitarian crises have been rigorously tested, and most studied interventions focused on posttraumatic stress disorder. Beyond posttraumatic stress disorder, individuals may have a range of problems including depression, anxiety, and not being able to do daily tasks necessary for survival and recovery. However, interventions are often limited since they tend to target only a single outcome, are usually of longer duration (8-16 sessions) or require professionals.

In low resourced settings interventions need to be short of duration, and be carried out by lay people in the communities to make them sustainable and feasible to implement on a broader scale. World Health Organization aims to develop a range of low-intensity scale-able psychological interventions that address these issues, as part of its mental health Gap Action Program. As a first step a simplified psychological intervention Problem Management Plus (PM+) has been developed. It has 4 core features that make the intervention suitable for low resourced setting exposed to adversities. First, it is brief intervention (5-sessions), delivered individually or in groups; second, it can be delivered by paraprofessionals (high school graduates with no mental health experience), using the principle of task shifting/ task sharing; third, it is designed as a trans- diagnostic intervention, addressing a range of client identified emotional (e.g. depression, anxiety, traumatic stress, general stress) and practical problems; fourth, it is designed for people in low-income country communities affected by any kind of adversity (e.g. violence, disasters), not just focusing on a single kind of adversity. Recent PM+ trails in Pakistan and Kenya have indicated PM+ to be effective in diminishing depression and anxiety and improving people's functioning and self- selected, culturally relevant outcomes. Group PM+ has been piloted in a district in Nepal, which was affected by the 2015 earthquakes. The pilot was conducted to gather information about the feasibility, safety and delivery of the intervention in the Nepali community settings; and to identify issues around training, supervision and outcomes measures. The pilot trial was successful in terms of acceptability and feasibility and detecting possible problems of compliance, delivery of the intervention, recruitment and retention. The current definitive study will evaluate the effectiveness of Group PM+ in Nepal through a pragmatic cluster randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. score YES to heart-mind problems on heart-mind screener
2. score >16 on World Health Organization Disability Assessment Scale

Exclusion Criteria:

1. Presence of a severe mental disorder (e.g., psychosis)
2. Alcohol use disorder (score >16 on the alcohol use disorders identification test (AUDIT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported gender
Enrollment: 611 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
General psychological distress - General Health Questionnaire | 20-weeks after baseline
  12-item measure of general psychological distress, validated in Nepal

SECONDARY OUTCOMES:
Daily functioning - World Health Organization Disability Assessment Scale | 20-weeks after baseline
  12-item assessment ability to engage in daily activities, previously used in numerous studies in Nepal
Depression - Patient Health Questionnaire | 20-weeks after baseline
  9-item measure of depression symptoms, culturally and clinically validated in Nepal
Posttraumatic Stress Disorder - Posttraumatic Stress Disorder Checklist | 20-weeks after baseline
  8-tem measure of post-traumatic stress symptoms validated for use in Nepal
Cultural idiom of psychological distress - Heart-Mind Screener | 20-weeks after baseline
  2-item locally develop psychological distress screener
Perceptions of support from family, friends, and others - Multidimensional Scale of Perceived Social Support | 20-weeks after baseline
  12-item assessment of perceptions of support from 3 sources: Family, Friends, and a Significant Other
Somatic symptom burden - Somatic Symptom Scale | 20-weeks after baseline
  8-item brief measure of somatic symptom burden

OTHER OUTCOMES:
Reducing Tension Checklist for Problem Management Plus Skills | 20-weeks after baseline
  10-item measure of behavioral and psychosocial skills related to coping mechanisms

CONTACTS AND LOCATIONS:
Overall Officials: Mark van Ommeren, PhD, Study Director — World Health Organization
Locations (1):
- Transcultural Psychosocial Organization (TPO) Nepal, Biratnagar, Morang, Nepal

IPD SHARING:
Plan to Share IPD: No
This will be shared for full trial.

REFERENCES:
- [Background] Bryant RA, Schafer A, Dawson KS, Anjuri D, Mulili C, Ndogoni L, Koyiet P, Sijbrandij M, Ulate J, Harper Shehadeh M, Hadzi-Pavlovic D, van Ommeren M. Effectiveness of a brief behavioural intervention on psychological distress among women with a history of gender-based violence in urban Kenya: A randomised clinical trial. PLoS Med. 2017 Aug 15;14(8):e1002371. doi: 10.1371/journal.pmed.1002371. eCollection 2017 Aug. PMID 28809935
- [Background] Khan MN, Hamdani SU, Chiumento A, Dawson K, Bryant RA, Sijbrandij M, Nazir H, Akhtar P, Masood A, Wang D, Wang E, Uddin I, van Ommeren M, Rahman A. Evaluating feasibility and acceptability of a group WHO trans-diagnostic intervention for women with common mental disorders in rural Pakistan: a cluster randomised controlled feasibility trial. Epidemiol Psychiatr Sci. 2019 Feb;28(1):77-87. doi: 10.1017/S2045796017000336. Epub 2017 Jul 10. PMID 28689511
- [Background] Hamdani SU, Ahmed Z, Sijbrandij M, Nazir H, Masood A, Akhtar P, Amin H, Bryant RA, Dawson K, van Ommeren M, Rahman A, Minhas FA. Problem Management Plus (PM+) in the management of common mental disorders in a specialized mental healthcare facility in Pakistan; study protocol for a randomized controlled trial. Int J Ment Health Syst. 2017 Jun 8;11:40. doi: 10.1186/s13033-017-0147-1. eCollection 2017. PMID 28603552
- [Background] Chiumento A, Hamdani SU, Khan MN, Dawson K, Bryant RA, Sijbrandij M, Nazir H, Akhtar P, Masood A, Wang D, van Ommeren M, Rahman A. Evaluating effectiveness and cost-effectiveness of a group psychological intervention using cognitive behavioural strategies for women with common mental disorders in conflict-affected rural Pakistan: study protocol for a randomised controlled trial. Trials. 2017 Apr 26;18(1):190. doi: 10.1186/s13063-017-1905-8. PMID 28441974
- [Background] Dawson KS, Schafer A, Anjuri D, Ndogoni L, Musyoki C, Sijbrandij M, van Ommeren M, Bryant RA. Feasibility trial of a scalable psychological intervention for women affected by urban adversity and gender-based violence in Nairobi. BMC Psychiatry. 2016 Nov 18;16(1):410. doi: 10.1186/s12888-016-1117-x. PMID 27863515
- [Background] Rahman A, Riaz N, Dawson KS, Usman Hamdani S, Chiumento A, Sijbrandij M, Minhas F, Bryant RA, Saeed K, van Ommeren M, Farooq S. Problem Management Plus (PM+): pilot trial of a WHO transdiagnostic psychological intervention in conflict-affected Pakistan. World Psychiatry. 2016 Jun;15(2):182-3. doi: 10.1002/wps.20312. No abstract available. PMID 27265713
- [Background] Sijbrandij M, Bryant RA, Schafer A, Dawson KS, Anjuri D, Ndogoni L, Ulate J, Hamdani SU, van Ommeren M. Problem Management Plus (PM+) in the treatment of common mental disorders in women affected by gender-based violence and urban adversity in Kenya; study protocol for a randomized controlled trial. Int J Ment Health Syst. 2016 May 31;10:44. doi: 10.1186/s13033-016-0075-5. eCollection 2016. PMID 27252778
- [Background] Sijbrandij M, Farooq S, Bryant RA, Dawson K, Hamdani SU, Chiumento A, Minhas F, Saeed K, Rahman A, van Ommeren M. Problem Management Plus (PM+) for common mental disorders in a humanitarian setting in Pakistan; study protocol for a randomised controlled trial (RCT). BMC Psychiatry. 2015 Oct 1;15:232. doi: 10.1186/s12888-015-0602-y. PMID 26428314
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Derived] Jordans MJD, Kohrt BA, Sangraula M, Turner EL, Wang X, Shrestha P, Ghimire R, Van't Hof E, Bryant RA, Dawson KS, Marahatta K, Luitel NP, van Ommeren M. Effectiveness of Group Problem Management Plus, a brief psychological intervention for adults affected by humanitarian disasters in Nepal: A cluster randomized controlled trial. PLoS Med. 2021 Jun 17;18(6):e1003621. doi: 10.1371/journal.pmed.1003621. eCollection 2021 Jun. PMID 34138875
- [Derived] Van't Hof E, Sangraula M, Luitel NP, Turner EL, Marahatta K, van Ommeren M, Shrestha P, Bryant R, Kohrt BA, Jordans MJD. Effectiveness of Group Problem Management Plus (Group-PM+) for adults affected by humanitarian crises in Nepal: study protocol for a cluster randomized controlled trial. Trials. 2020 Apr 19;21(1):343. doi: 10.1186/s13063-020-04263-9. PMID 32307009